CLINICAL TRIAL: NCT06559683
Title: Comparison of Maximum Extension of Sensory Assessment Following Superficial and Deep Parasternal Intercostal Plane Blocks
Brief Title: Comparison of Sensory Analysis After Superficial and Deep Parasternal Intercostal Plane Blocks
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, associate professor, Ondokuz Mayıs University
Other Study IDs: SensoryParasternal
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative
Keywords: analgesia; pain Management; sensory assessment
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep Parasternal: Patients scheduled for open-heart surgery will receive a deep parasternal intercostal plane block preoperatively, and sensory block status will be evaluated 30 minutes later using small ice tubes.
  Interventions: Other: Sensory Assessment
- Superficial Parasternal: Patients scheduled for open-heart surgery will receive a superficial parasternal intercostal plane block preoperatively, and sensory block status will be evaluated 30 minutes later using small ice tubes.
  Interventions: Other: Sensory Assessment

INTERVENTIONS:
Other: Sensory Assessment — Patients scheduled for open-heart surgery will receive a deep/superficial parasternal intercostal plane block preoperatively, and sensory block status will be evaluated after 30 minutes.

SUMMARY:
Postoperative pain following cardiac surgery is a common issue that can negatively impact patients' quality of life. Effective perioperative pain management is crucial to improving patient outcomes. Pain is typically most intense during the first two postoperative days, and inadequate management can lead to chronic pain, further diminishing quality of life. Recent advances in ultrasound-guided regional anesthesia, including superficial and deep parasternal intercostal plane blocks, have enhanced acute pain control. These blocks aim to provide analgesia by targeting the anterior cutaneous branches of the T2-6 thoracic nerves. While their efficacy is recognized, sensory evaluation and dermatomal analysis remain unexplored. Cadaver studies suggest that the deep block may cover more parasternal space than the superficial block.

DETAILED DESCRIPTION:
This observational study evaluates sensory blocks in patients undergoing open-heart surgery who receive superficial or deep parasternal intercostal plane blocks. Sensory assessment, conducted by a blinded researcher 30 minutes post-block, involves applying small ice tubes with cold sensations categorized as Normal, Reduced, or No cold. A successful block is defined as the loss or reduction of cold sensitivity, while normal cold sensation indicates block failure. Assessments start at the midline, moving laterally to the anterior axillary line. Marked areas are digitally analyzed. Block regression is evaluated at 12 and 24 hours post-procedure using the same cold assessment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo effective open heart surgery with median sternotomy
* Patients who have undergone superficial or deep parasternal intercostal plane block

Exclusion Criteria:

* Patients with severe psychiatric illnesses such as psychosis or dementia that would prevent communication with the patient
* Patients who do not want to participate in the study
* Redo surgeries
* Patients whose block is considered unsuccessful with the cold application test at the 30th minute
* Patients who cannot be extubated 12 hours post-block.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for median sternotomy as part of open-heart surgery and who have received either a superficial or deep parasternal intercostal plane block will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Extent of Sensory Blockade Measured by Cold Sensation Testing Across the Anterior Chest Wall Following Deep and Superficial Parasternal Intercostal Plane Blocks. | 30 minutes after the blocks
  Participants will undergo sensory assessment using standardized cold sensation test at 30 minutes post-block to evaluate the maximum sensory blockade. The data will be recorded as the area of sensory loss (in cm) along the anterior chest wall, and the results will be aggregated to report the maximum area of sensory blockade achieved for both deep and superficial blocks. Cold sensation will be categorized as Normal Cold, Reduced Cold, or No Cold Sensation. A successful block is defined as a complete loss or reduction of cold sensitivity.

SECONDARY OUTCOMES:
Regression of Sensory Blockade at 12 and 24 Hours Post-Block | Postoperative Day 1
  Block regression will be evaluated at 12 and 24 hours after block administration using cold sensation testing with ice tubes. The cold sensation will be categorized as Normal Cold, Reduced Cold, or No Cold Sensation. Participants who report Normal Cold sensation will be considered to have experienced block regression.
Opioid Consumption | Postoperative Day 1
  Opioid consumption at 12, and 24 hours after block administration will be measured by IV patient controlled analgesia.
Acute pain scores | Postoperative Day 1
  Pain status at rest and while coughing will be assessed by Numeric Rating Scale (NRS) scores at 12, and 24 hours after block administration.The NRS is an 11-point numeric scale which ranges from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)